CLINICAL TRIAL: NCT04401579
Title: A Multicenter, Adaptive, Randomized Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for the Treatment of COVID-19 in Hospitalized Adults (ACTT-2)
Brief Title: Adaptive COVID-19 Treatment Trial 2 (ACTT-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-0006 ACTT-2
Record Dates: First submitted 2020-05-22; First posted 2020-05-26 (Actual); Results first posted 2021-04-26 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Adaptive; COVID-19; Efficacy; Multicenter; novel coronavirus; Safety
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remdesivir plus Baricitinib (Experimental): 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10-day total course and 4 mg (2 tablets of 2 mg) of Baricitinib administered orally daily for the duration of the hospitalization up to a 14-day total course.
  Interventions: Drug: Remdesivir; Drug: Baricitinib
- Remdesivir plus Placebo (Placebo Comparator): 200 mg of Remdesivir administered intravenously on Day 1, followed by a 100 mg once-daily maintenance dose of Remdesivir while hospitalized for up to a 10-day total course and 4 mg (2 tablets of 2 mg) of Baricitinib Placebo administered orally daily for the duration of the hospitalization up to a 14-day total course.
  Interventions: Other: Placebo; Drug: Remdesivir

INTERVENTIONS:
Other: Placebo — The matching Baricitinib placebo contains lactose monohydrate, microcrystalline cellulose, croscarmellose sodium, and magnesium stearate. The coating for the placebo tablet is identical to that of the corresponding active tablet.
  Arms: Remdesivir plus Placebo
Drug: Remdesivir — Drug Remdesivir is a single diastereomer monophosphoramidate prodrug designed for the intracellular delivery of a modified adenine nucleoside analog GS-441524. In addition to the active ingredient, the lyophilized formulation of Remdesivir contains the following inactive ingredients: water for injection, sulfobutylether beta-cyclodextrin sodium (SBECD), and hydrochloric acid and/or sodium hydroxide.
Drug: Baricitinib — Baricitinib is a Janus kinase (JAK) inhibitor with the chemical name [1-(ethylsulfonyl)-3-(4-(7Hpyrrolo(2,3-d)pyrimidin-4-yl)-1H-pyrazol-1-yl)azetidin-3-yl]acetonitrile Each tablet contains 2 mg of baricitinib and the following inactive ingredients: croscarmellose sodium, magnesium stearate, mannitol, microcrystalline cellulose, ferric oxide, lecithin (soya), polyethylene glycol, polyvinyl alcohol, talc and titanium dioxide.
  Arms: Remdesivir plus Baricitinib

SUMMARY:
ACTT-2 will evaluate the combination of baricitinib and remdesivir compared to remdesivir alone. Subjects will be assessed daily while hospitalized. If the subjects are discharged from the hospital, they will have a study visit at Days 15, 22, and 29. For discharged subjects, it is preferred that the Day 15 and 29 visits are in person to obtain safety laboratory tests and oropharyngeal (OP) swab and blood (serum only) samples for secondary research as well as clinical outcome data. However, infection control or other restrictions may limit the ability of the subject to return to the clinic. In this case, these visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and is conducted by phone. The primary outcome is time to recovery by Day 29.

DETAILED DESCRIPTION:
This study is an adaptive randomized double-blind placebo-controlled trial to evaluate the safety and efficacy of novel therapeutic agents in hospitalized adults diagnosed with COVID-19. The study is a multicenter trial that will be conducted in up to approximately 100 sites globally. The study will compare different investigational therapeutic agents to a control arm. New arms can be introduced according to scientific and public health needs. There will be interim monitoring to allow early stopping for futility, efficacy, or safety. If one therapy proves to be efficacious, then this treatment may become the control arm for comparison(s) with new experimental treatment(s). Any such change would be accompanied by an updated sample size. This adaptive platform is used to rapidly evaluate different therapeutics in a population of those hospitalized with moderate to severe COVID-19. The platform will provide a common framework sharing a similar population, design, endpoints, and safety oversight. New stages with new therapeutics can be introduced. One independent Data and Safety Monitoring Board (DSMB) will actively monitor interim data in all stages to make recommendations about early study closure or changes to study arms.

ACTT-2 will evaluate the combination of baricitinib and remdesivir compared to remdesivir alone. Subjects will be assessed daily while hospitalized. If the subjects are discharged from the hospital, they will have a study visit at Days 15, 22, and 29. For discharged subjects, it is preferred that the Day 15 and 29 visits are in person to obtain safety laboratory tests and oropharyngeal (OP) swab and blood (serum only) samples for secondary research as well as clinical outcome data. However, infection control or other restrictions may limit the ability of the subject to return to the clinic. In this case, these visits may be conducted by phone, and only clinical data will be obtained. The Day 22 visit does not have laboratory tests or collection of samples and is conducted by phone.

All subjects will undergo a series of efficacy, safety, and laboratory assessments. Safety laboratory tests and blood (serum and plasma) research samples and oropharyngeal (OP) swabs will be obtained on Days 1 (prior to infusion) and Days 3, 5, 8, and 11 (while hospitalized). OP swabs and blood (serum only) plus safety laboratory tests will be collected on Day 15 and 29 (if the subject attends an in-person visit or are still hospitalized).

The primary outcome is time to recovery by Day 29. A key secondary outcome evaluates treatment-related improvements in the 8-point ordinal scale at Day 15. Each stage may prioritize different secondary endpoints for the purpose of multiple comparison analyses.

Contacts:

20-0006 Central Contact

Telephone: 1 (301) 7617948

Email: DMIDClinicalTrials@niaid.nih.gov

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to a hospital with symptoms suggestive of COVID-19.
2. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
3. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
4. Male or non-pregnant female adult > / = 18 years of age at time of enrollment.
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by polymerase chain reaction (PCR) or other commercial or public health assay in any specimen, as documented by either of the following:

   * PCR positive in sample collected < 72 hours prior to randomization; OR
   * PCR positive in sample collected >/= 72 hours prior to randomization, documented inability to obtain a repeat sample (e.g. due to lack of testing supplies, limited testing capacity, results taking >24 hours, etc.) AND progressive disease suggestive of ongoing SARS-CoV-2 infection.
6. Illness of any duration, and at least one of the following:

   * Radiographic infiltrates by imaging (chest x-ray, CT scan, etc.), OR
   * SpO2 < / = 94% on room air, OR
   * Requiring supplemental oxygen, OR
   * Requiring mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
7. Women of childbearing potential must agree to either abstinence or use at least one primary form of contraception not including hormonal contraception from the time of screening through Day 29.
8. Agrees to not participate in another clinical trial for the treatment of COVID-19 through Day 29.

Exclusion Criteria:

1. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
2. Estimated glomerular filtration rate (eGFR) < 30 ml/min or patient is receiving hemodialysis or hemofiltration at time of screening.
3. Neutropenia (absolute neutrophil count <1000 cells/microliter) (<1.0 x 103/microliter or <1.0 GI/L).
4. Lymphopenia (absolute lymphocyte count <200 cells/microliter) (<0.20 x 103/microliter or <0.20 GI/L)
5. Pregnancy or breast feeding.
6. Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 72 hours.
7. Allergy to any study medication.
8. Received three or more doses of remdesivir, including the loading dose, outside of the study under the EUA (or similar mechanism) for COVID-19.
9. Received convalescent plasma or intravenous immunoglobulin [IVIg]) for COVID-19, the current illness for which they are being enrolled.
10. Received small molecule tyrosine kinase inhibitors (e.g. baricitinib, imatibib, genfinitib), in the 1 week prior to screening
11. Received monoclonal antibodies targeting cytokines (e.g., TNF inhibitors, anti-interleukin-1 [IL-1], anti-IL-6 [tocilizumab or sarilumab]), or T-cells (e.g., abatacept) in the 4 weeks prior to screening.
12. Received monoclonal antibodies targeting B-cell (e.g., rituximab, and including any targeting multiple cell lines including B-cells) in the 3 months prior to screening.
13. Received other immunosuppressants in the 4 weeks prior to screening and in the judgement of the investigator, the risk of immunosuppression with baricitinib is larger than the risk of COVID-19.
14. Received >/= 20 mg/day of prednisone or equivalent for >/=14 consecutive days in the 4 weeks prior to screening.
15. Use of probenecid that cannot be discontinued at study enrollment.
16. Have diagnosis of current active tuberculosis (TB) or, if known, latent TB treated for less than 4 weeks with appropriate anti-tuberculosis therapy per local guidelines (by history only, no screening required).
17. Suspected serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking investigational product.
18. Have received any live vaccine (that is, live attenuated) within 4 weeks before screening, or intend to receive a live vaccine (or live attenuated) during the study. Note: Use of non-live (inactivated) vaccinations is allowed for all subjects.
19. Have a history of VTE (deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 12 weeks prior to screening or have a history of recurrent (>1) VTE (DVT/PE).
20. Immunocompromised patients, patients with a chronic medical condition, or those taking a medication that cannot be discontinued at enrollment, who, in the judgment of PI, are at increased risk for serious infections or other safety concerns given the study products.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1033 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (71):
- United States (53):
  - University of Alabama at Birmingham School of Medicine - Infectious Disease, Birmingham, Alabama
  - University of California San Diego Health - Jacobs Medical Center, La Jolla, California
  - University of California Los Angeles Medical Center - Westwood Clinic, Los Angeles, California
  - University of California Irvine Medical Center - Infectious Disease, Orange, California
  - VA Palo Alto Health Care System - Infectious Diseases, Palo Alto, California
  - Stanford University - Stanford Hospital and Clinics - Pediatrics - Infectious Diseases, Palo Alto, California
  - University of California Davis Medical Center - Internal Medicine - Infectious Disease, Sacramento, California
  - Naval Medical Center San Diego - Infectious Disease Clinic, San Diego, California
  - University of California San Francisco - Zuckerberg San Francisco General Hospital - Division of Human Immunodeficiency Virus, Infectious Disease, and Global Medicine, San Francisco, California
  - Cedars Sinai Medical Center, West Hollywood, California
  - Eastern Colorado Health Care System, Aurora, Colorado
  - Denver Health Division of Hospital Medicine - Main Campus, Denver, Colorado
  - Georgetown University Medical Center - Division of Infectious Diseases, Washington D.C., District of Columbia
  - University of Florida Health - Shands Hospital - Division of Infectious Diseases and Global Medicine, Gainesville, Florida
  - University of Miami Miller School of Medicine - Infectious Diseases, Miami, Florida
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - Atlanta VA Medical Center - Infectious Diseases Clinic, Decatur, Georgia
  - Northwestern Hospital - Infectious Disease, Chicago, Illinois
  - University of Illinois at Chicago College of Medicine - Division of Infectious Diseases, Chicago, Illinois
  - Indiana University School of Medicine - Infectious Diseases, Indianapolis, Indiana
  - Ochsner Medical Center - Kenner - Department of Infectious Diseases, Kenner, Louisiana
  - Southeast Louisiana Veterans Health Care System (SLVHCS) - Section of Infectious Diseases, New Orleans, Louisiana
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Johns Hopkins Hospital - Medicine - Infectious Diseases, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - National Institutes of Health - Clinical Center, National Institute of Allergy and Infectious Diseases Laboratory Of Immunoregulation, Clinical Research Section, Bethesda, Maryland
  - Massachusetts General Hospital - Infectious Diseases, Boston, Massachusetts
  - University of Massachusetts Medical School - Infectious Diseases and Immunology, Worcester, Massachusetts
  - University of Minnesota Medical Center, Fairview - Infectious Diseases and International Medicine, Minneapolis, Minnesota
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - University of Nebraska Medical Center - Infectious Diseases, Omaha, Nebraska
  - University of New Mexico Clinical and Translational Science Center, Albuquerque, New Mexico
  - New York University School of Medicine - Langone Medical Center - Microbiology - Parasitology, New York, New York
  - University of Rochester Medical Center - Vaccine Research Unit, Rochester, New York
  - Montefiore Medical Center - Infectious Diseases, The Bronx, New York
  - Duke Human Vaccine Institute - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Womack Army Medical Center - Pulmonary and Respiratory Services, Fort Bragg, North Carolina
  - Kaiser Permanente Northwest - Center for Health Research, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center - Division of Infectious Diseases, Hershey, Pennsylvania
  - University of Pennsylvania Perelman School of Medicine - Penn Institute for Immunology, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center - Infectious Diseases, Nashville, Tennessee
  - Baylor Scott & White Health - Baylor University Medical Center - North Texas Infectious Disease Consultants, Dallas, Texas
  - University of Texas Southwestern Medical Center - Internal Medicine - Infectious Diseases, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch - Division of Infectious Disease, Galveston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - University of Texas Health Science Center at San Antonio - Infectious Diseases, San Antonio, Texas
  - University of Utah - Infectious Diseases, Salt Lake City, Utah
  - University of Virginia - Acute Care Surgery, Charlottesville, Virginia
  - Naval Medical Center Portsmouth - Infectious Disease Division, Portsmouth, Virginia
  - EvergreenHealth Infectious Disease Service, Kirkland, Washington
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Madigan Army Medical Center - Infectious Disease Clinic, Tacoma, Washington
- University of Copenhagen - Centre of Excellence for Health, Immunity and Infections (CHIP) - Department of Infectious Diseases, Copenhagen, Denmark
- National Center for Global Health and Medicine Hospital - Disease Control and Prevention Center, Tokyo, Japan
- Mexico (2):
  - Instituto Nacional de Ciencias Medicas y Nutrición Salvador Zubirán - Departamento de Infectologia, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias (INER) - Ismael Cosío Villegas, Mexico City
- Singapore (4):
  - National University Health System - Division of Infectious Diseases, Singapore
  - National Centre for Infectious Diseases (NCID), Singapore
  - Changi General Hospital - Clinical Trials and Research Unit (CTRU), Singapore
  - Ng Teng Fong General Hospital - Infectious Disease Service, Singapore
- South Korea (2):
  - Seoul National University Bundang Hospital - Division of Infectious Diseases, Bundang-gu Seongnam-si
  - Seoul National University Hospital, Seoul
- Spain (3):
  - Hospital Clinic Barcelona, Servicio de Salud Internacional, Barcelona, Catalonia
  - Hospital Germans Trias i Pujol - Servei Malalties Infeccioses, Barcelona, Catalonia
  - Hospital Clinico San Carlos - Enfermedades Infecciosas, Madrid
- United Kingdom (5):
  - Royal Sussex County Hospital - Department of Intensive Care Medicine, Brighton
  - Saint Thomas' Hospital - Directorate of Infection, City of London
  - St. James's University Hospital - Infectious Diseases, Leeds
  - Royal Victoria Infirmary - Department of Infectious Diseases, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Paules CI, Wang J, Tomashek KM, Bonnett T, Singh K, Marconi VC, Davey RT Jr, Lye DC, Dodd LE, Yang OO, Benson CA, Deye GA, Doernberg SB, Hynes NA, Grossberg R, Wolfe CR, Nayak SU, Short WR, Voell J, Potter GE, Rapaka RR. A Risk Profile Using Simple Hematologic Parameters to Assess Benefits From Baricitinib in Patients Hospitalized With COVID-19: A Post Hoc Analysis of the Adaptive COVID-19 Treatment Trial-2. Ann Intern Med. 2024 Mar;177(3):343-352. doi: 10.7326/M23-2593. Epub 2024 Feb 27. PMID 38408357
- [Derived] Potter GE, Bonnett T, Rubenstein K, Lindholm DA, Rapaka RR, Doernberg SB, Lye DC, Mularski RA, Hynes NA, Kline S, Paules CI, Wolfe CR, Frank MG, Rouphael NG, Deye GA, Sweeney DA, Colombo RE, Davey RT Jr, Mehta AK, Whitaker JA, Castro JG, Amin AN, Colombo CJ, Levine CB, Jain MK, Maves RC, Marconi VC, Grossberg R, Hozayen S, Burgess TH, Atmar RL, Ganesan A, Gomez CA, Benson CA, Lopez de Castilla D, Ahuja N, George SL, Nayak SU, Cohen SH, Lalani T, Short WR, Erdmann N, Tomashek KM, Tebas P. Temporal Improvements in COVID-19 Outcomes for Hospitalized Adults: A Post Hoc Observational Study of Remdesivir Group Participants in the Adaptive COVID-19 Treatment Trial. Ann Intern Med. 2022 Dec;175(12):1716-1727. doi: 10.7326/M22-2116. Epub 2022 Nov 29. PMID 36442063
- [Derived] Kramer A, Prinz C, Fichtner F, Fischer AL, Thieme V, Grundeis F, Spagl M, Seeber C, Piechotta V, Metzendorf MI, Golinski M, Moerer O, Stephani C, Mikolajewska A, Kluge S, Stegemann M, Laudi S, Skoetz N. Janus kinase inhibitors for the treatment of COVID-19. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD015209. doi: 10.1002/14651858.CD015209. PMID 35695334
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Kalil AC, Patterson TF, Mehta AK, Tomashek KM, Wolfe CR, Ghazaryan V, Marconi VC, Ruiz-Palacios GM, Hsieh L, Kline S, Tapson V, Iovine NM, Jain MK, Sweeney DA, El Sahly HM, Branche AR, Regalado Pineda J, Lye DC, Sandkovsky U, Luetkemeyer AF, Cohen SH, Finberg RW, Jackson PEH, Taiwo B, Paules CI, Arguinchona H, Erdmann N, Ahuja N, Frank M, Oh MD, Kim ES, Tan SY, Mularski RA, Nielsen H, Ponce PO, Taylor BS, Larson L, Rouphael NG, Saklawi Y, Cantos VD, Ko ER, Engemann JJ, Amin AN, Watanabe M, Billings J, Elie MC, Davey RT, Burgess TH, Ferreira J, Green M, Makowski M, Cardoso A, de Bono S, Bonnett T, Proschan M, Deye GA, Dempsey W, Nayak SU, Dodd LE, Beigel JH; ACTT-2 Study Group Members. Baricitinib plus Remdesivir for Hospitalized Adults with Covid-19. N Engl J Med. 2021 Mar 4;384(9):795-807. doi: 10.1056/NEJMoa2031994. Epub 2020 Dec 11. PMID 33306283
- [Derived] Azzi Y, Bartash R, Scalea J, Loarte-Campos P, Akalin E. COVID-19 and Solid Organ Transplantation: A Review Article. Transplantation. 2021 Jan 1;105(1):37-55. doi: 10.1097/TP.0000000000003523. PMID 33148977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the participating sites from those admitted with symptoms of COVID-19 confirmed by PCR. Enrollment occurred between 08May2020 and 01Jul2020.
Period: Overall Study
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Started | 515 | 518
Treated | 507 | 509
Completed | 431 | 408
Not Completed | 84 | 110
Not completed — Death | 23 | 36
Not completed — Lost to Follow-up | 40 | 41
Not completed — Withdrawal by Subject | 8 | 16
Not completed — Physician Decision | 1 | 2
Not completed — Became ineligible after enrollment | 1 | 1
Not completed — Enrolled but treatment not administered | 7 | 9
Not completed — Adverse Event | 2 | 1
Not completed — Scheduling error | 1 | 2
Not completed — Transferred to another hospital | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo | Total
Number analyzed (Participants) | 515 | 518 | 1033
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 368 | 360 | 728
  >=65 years | 147 | 158 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (15.4) | 55.8 (16.0) | 55.4 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 185 | 381
  Male | 319 | 333 | 652
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 263 | 268 | 531
  Not Hispanic or Latino | 246 | 240 | 486
  Unknown or Not Reported | 6 | 10 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 8 | 10
  Asian | 49 | 52 | 101
  Native Hawaiian or Other Pacific Islander | 4 | 7 | 11
  Black or African American | 77 | 79 | 156
  White | 251 | 245 | 496
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 132 | 127 | 259
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 11 | 11 | 22
  Singapore | 22 | 22 | 44
  United States | 441 | 444 | 885
  Japan | 0 | 1 | 1
  Denmark | 4 | 5 | 9
  Mexico | 35 | 33 | 68
  United Kingdom | 0 | 1 | 1
  Spain | 2 | 1 | 3
Disease severity [Count of Participants; unit: Participants] — Severe disease was defined as hospitalized, requiring extracorporeal membrane oxygenation (ECMO), invasive or non-invasive ventilation, or high flow oxygen Moderate disease was defined as hospitalized, requiring supplemental oxygen or not requiring supplemental oxygen.
  Disease severity was as defined at the time or randomization.
  Participants
    Severe Disease Severity | 176 | 191 | 367
    Moderate Disease Severity | 339 | 327 | 666

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery
Description: Day of recovery is defined as the first day on which the subject satisfies one of the following three categories from the ordinal scale: 1) Not hospitalized, no limitations on activities; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 3) Hospitalized, not requiring supplemental oxygen and no longer requires ongoing medical care.
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
Days | 7.0 [6.0 to 8.0] | 8.0 [7.0 to 9.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; Test type: Superiority; p = 0.047, Log Rank; Cox Proportional Hazard = 1.15, 95% CI 2-sided [1.00 to 1.31]

2. Secondary Outcome: Change From Baseline in Alanine Transaminase (ALT)
Description: Blood to evaluate ALT was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: The safety population includes all treated participants with available data at baseline and the post baseline assessment point, analyzed as treated.
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 491 | 491
Units/Liter (U/L)
  Day 3 | 3.3 (37.1) | 2.0 (30.1)
  Day 5: number analyzed (Participants) | 407 | 406
  Day 5 | 16.8 (104.4) | 8.8 (40.9)
  Day 8: number analyzed (Participants) | 268 | 284
  Day 8 | 7.9 (45.2) | 7.8 (46.9)
  Day 11: number analyzed (Participants) | 187 | 201
  Day 11 | 0.0 (37.5) | 7.3 (70.2)
  Day 15: number analyzed (Participants) | 250 | 270
  Day 15 | 5.0 (61.5) | 3.9 (55.1)
  Day 29: number analyzed (Participants) | 256 | 255
  Day 29 | -5.4 (43.0) | 2.3 (116.1)

3. Secondary Outcome: Change From Baseline in Aspartate Transaminase (AST)
Description: Blood to evaluate AST was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 486 | 487
Units/Liter (U/L)
  Day 3 | 3.1 (72.4) | 2.4 (126.4)
  Day 5: number analyzed (Participants) | 404 | 403
  Day 5 | 27.4 (413.1) | 2.8 (48.3)
  Day 8: number analyzed (Participants) | 265 | 282
  Day 8 | -5.6 (38.4) | -4.3 (42.3)
  Day 11: number analyzed (Participants) | 185 | 200
  Day 11 | -10.6 (46.4) | 6.4 (208.3)
  Day 15: number analyzed (Participants) | 246 | 266
  Day 15 | -6.0 (110.1) | -3.9 (91.0)
  Day 29: number analyzed (Participants) | 251 | 251
  Day 29 | -17.1 (46.7) | 2.4 (291.1)

4. Secondary Outcome: Change From Baseline in Creatinine
Description: Blood to evaluate serum creatinine was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: milligrams/deciliter (mg/dL)
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 494 | 495
milligrams/deciliter (mg/dL)
  Day 3 | -0.036 (0.465) | -0.019 (0.362)
  Day 5: number analyzed (Participants) | 412 | 410
  Day 5 | -0.078 (0.475) | 0.001 (0.556)
  Day 8: number analyzed (Participants) | 270 | 285
  Day 8 | -0.082 (0.570) | 0.129 (0.958)
  Day 11: number analyzed (Participants) | 190 | 202
  Day 11 | -0.055 (0.798) | 0.194 (1.037)
  Day 15: number analyzed (Participants) | 254 | 273
  Day 15 | -0.042 (0.714) | 0.094 (0.662)
  Day 29: number analyzed (Participants) | 260 | 257
  Day 29 | -0.034 (0.678) | 0.033 (0.511)

5. Secondary Outcome: Change From Baseline in Glucose
Description: Blood to evaluate serum glucose was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 493 | 493
mg/dL
  Day 3 | -17.1 (56.4) | -6.0 (54.0)
  Day 5: number analyzed (Participants) | 412 | 409
  Day 5 | -15.9 (59.7) | -1.6 (58.4)
  Day 8: number analyzed (Participants) | 270 | 284
  Day 8 | -16.8 (78.9) | 5.0 (73.7)
  Day 11: number analyzed (Participants) | 190 | 203
  Day 11 | -8.1 (72.3) | 1.2 (66.2)
  Day 15: number analyzed (Participants) | 252 | 271
  Day 15 | -11.1 (69.8) | 0.8 (68.3)
  Day 29: number analyzed (Participants) | 257 | 256
  Day 29 | -4.6 (66.5) | -2.2 (60.3)

6. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Blood to evaluate hemoglobin was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams/deciliter (g/dL)
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 493 | 494
grams/deciliter (g/dL)
  Day 3 | -0.46 (1.05) | -0.34 (1.51)
  Day 5: number analyzed (Participants) | 410 | 409
  Day 5 | -0.62 (1.23) | -0.64 (1.13)
  Day 8: number analyzed (Participants) | 270 | 284
  Day 8 | -0.93 (1.61) | -1.08 (1.47)
  Day 11: number analyzed (Participants) | 189 | 199
  Day 11 | -1.29 (1.85) | -1.62 (1.88)
  Day 15: number analyzed (Participants) | 253 | 267
  Day 15 | -0.96 (1.87) | -1.12 (2.38)
  Day 29: number analyzed (Participants) | 260 | 254
  Day 29 | -0.54 (1.87) | -0.77 (2.25)

7. Secondary Outcome: Change From Baseline in Platelets
Description: Blood to evaluate platelets was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 493 | 494
10^9 cells/liter
  Day 3 | 55.9 (54.0) | 52.6 (51.6)
  Day 5: number analyzed (Participants) | 410 | 409
  Day 5 | 116.6 (87.8) | 106.1 (86.9)
  Day 8: number analyzed (Participants) | 269 | 284
  Day 8 | 197.9 (137.4) | 158.9 (128.5)
  Day 11: number analyzed (Participants) | 189 | 199
  Day 11 | 229.9 (156.0) | 145.7 (146.4)
  Day 15: number analyzed (Participants) | 252 | 267
  Day 15 | 175.9 (158.8) | 111.6 (134.9)
  Day 29: number analyzed (Participants) | 260 | 254
  Day 29 | 16.5 (95.8) | 36.9 (107.9)

8. Secondary Outcome: Change From Baseline in Prothrombin International Normalized Ratio (INR)
Description: Blood to evaluate INR was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 447 | 439
ratio
  Day 3 | -0.03 (1.13) | 0.05 (0.59)
  Day 5: number analyzed (Participants) | 360 | 370
  Day 5 | 0.02 (1.25) | 0.08 (0.65)
  Day 8: number analyzed (Participants) | 244 | 250
  Day 8 | 0.01 (0.96) | 0.08 (0.98)
  Day 11: number analyzed (Participants) | 162 | 175
  Day 11 | 0.04 (0.65) | 0.03 (1.04)
  Day 15: number analyzed (Participants) | 222 | 241
  Day 15 | -0.04 (0.25) | -0.08 (0.91)
  Day 29: number analyzed (Participants) | 232 | 232
  Day 29 | -0.12 (0.55) | -0.03 (0.99)

9. Secondary Outcome: Change From Baseline in Total Bilirubin
Description: Blood to evaluate total bilirubin was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 490 | 491
mg/dL
  Day 3 | -0.06 (0.32) | -0.01 (0.43)
  Day 5: number analyzed (Participants) | 407 | 405
  Day 5 | -0.04 (0.37) | 0.01 (0.42)
  Day 8: number analyzed (Participants) | 268 | 284
  Day 8 | -0.06 (0.41) | 0.01 (0.66)
  Day 11: number analyzed (Participants) | 187 | 201
  Day 11 | -0.08 (0.43) | 0.08 (1.19)
  Day 15: number analyzed (Participants) | 250 | 270
  Day 15 | -0.10 (0.37) | 0.08 (1.20)
  Day 29: number analyzed (Participants) | 256 | 254
  Day 29 | -0.10 (0.36) | 0.01 (0.91)

10. Secondary Outcome: Change From Baseline in White Blood Cell Count (WBC)
Description: Blood to evaluate WBC was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 493 | 494
10^9 cells/liter
  Day 3 | -0.831 (3.020) | -0.037 (2.588)
  Day 5: number analyzed (Participants) | 410 | 409
  Day 5 | -0.276 (3.399) | 0.392 (3.238)
  Day 8: number analyzed (Participants) | 270 | 284
  Day 8 | 0.663 (4.006) | 1.606 (4.536)
  Day 11: number analyzed (Participants) | 189 | 199
  Day 11 | 1.869 (5.683) | 2.938 (5.419)
  Day 15: number analyzed (Participants) | 253 | 267
  Day 15 | 0.694 (5.125) | 2.162 (5.741)
  Day 29: number analyzed (Participants) | 260 | 254
  Day 29 | -0.364 (4.532) | 0.712 (4.176)

11. Secondary Outcome: Change From Baseline in Neutrophils
Description: BBlood to evaluate neutrophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 488 | 493
10^9 cells/liter
  Day 3 | -1.925 (6.234) | -0.333 (2.787)
  Day 5: number analyzed (Participants) | 408 | 404
  Day 5 | -1.334 (8.092) | -0.204 (3.630)
  Day 8: number analyzed (Participants) | 268 | 282
  Day 8 | -0.813 (9.695) | 1.139 (6.665)
  Day 11: number analyzed (Participants) | 186 | 196
  Day 11 | -0.046 (8.881) | 1.847 (5.152)
  Day 15: number analyzed (Participants) | 249 | 267
  Day 15 | -1.192 (7.844) | 1.414 (7.995)
  Day 29: number analyzed (Participants) | 257 | 253
  Day 29 | -1.708 (6.735) | -0.656 (4.205)

12. Secondary Outcome: Change From Baseline in Lymphocytes
Description: Blood to evaluate lymphocytes was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 488 | 493
10^9 cells/liter
  Day 3 | 0.503 (2.290) | 0.074 (3.844)
  Day 5: number analyzed (Participants) | 408 | 404
  Day 5 | 0.620 (2.540) | 0.205 (3.838)
  Day 8: number analyzed (Participants) | 268 | 282
  Day 8 | 0.515 (2.094) | 0.304 (1.366)
  Day 11: number analyzed (Participants) | 186 | 196
  Day 11 | 0.541 (1.204) | 0.409 (0.709)
  Day 15: number analyzed (Participants) | 249 | 267
  Day 15 | 0.687 (1.579) | 0.718 (1.684)
  Day 29: number analyzed (Participants) | 257 | 253
  Day 29 | 0.653 (1.293) | 0.927 (1.996)

13. Secondary Outcome: Change From Baseline in Monocytes
Description: Blood to evaluate monocytes was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 487 | 493
10^9 cells/liter
  Day 3 | 0.004 (0.810) | 0.062 (0.750)
  Day 5: number analyzed (Participants) | 408 | 404
  Day 5 | 0.094 (1.053) | 0.153 (1.013)
  Day 8: number analyzed (Participants) | 268 | 282
  Day 8 | 0.105 (0.948) | 0.279 (0.758)
  Day 11: number analyzed (Participants) | 186 | 196
  Day 11 | 0.210 (0.439) | 0.378 (0.512)
  Day 15: number analyzed (Participants) | 249 | 267
  Day 15 | 0.256 (0.591) | 0.329 (0.606)
  Day 29: number analyzed (Participants) | 257 | 253
  Day 29 | 0.108 (0.434) | 0.212 (0.745)

14. Secondary Outcome: Change From Baseline in Basophils
Description: Blood to evaluate basophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 483 | 492
10^9 cells/liter
  Day 3 | 0.000 (0.039) | 0.001 (0.050)
  Day 5: number analyzed (Participants) | 402 | 402
  Day 5 | 0.007 (0.070) | 0.006 (0.044)
  Day 8: number analyzed (Participants) | 265 | 281
  Day 8 | 0.011 (0.055) | 0.017 (0.075)
  Day 11: number analyzed (Participants) | 185 | 195
  Day 11 | 0.014 (0.063) | 0.022 (0.063)
  Day 15: number analyzed (Participants) | 247 | 265
  Day 15 | 0.026 (0.085) | 0.037 (0.104)
  Day 29: number analyzed (Participants) | 257 | 250
  Day 29 | 0.022 (0.045) | 0.036 (0.092)

15. Secondary Outcome: Change From Baseline in Eosinophils
Description: Blood to evaluate eosinophils was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 10^9 cells/liter
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 484 | 492
10^9 cells/liter
  Day 3 | 0.050 (0.135) | 0.039 (0.201)
  Day 5: number analyzed (Participants) | 405 | 403
  Day 5 | 0.104 (0.402) | 0.075 (0.257)
  Day 8: number analyzed (Participants) | 265 | 281
  Day 8 | 0.088 (0.126) | 0.086 (0.232)
  Day 11: number analyzed (Participants) | 185 | 195
  Day 11 | 0.078 (0.119) | 0.115 (0.299)
  Day 15: number analyzed (Participants) | 247 | 264
  Day 15 | 0.121 (0.231) | 0.109 (0.163)
  Day 29: number analyzed (Participants) | 257 | 251
  Day 29 | 0.192 (0.171) | 0.205 (0.267)

16. Secondary Outcome: Change in National Early Warning Score (NEWS) From Baseline
Description: The NEW score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness). The NEW Score is being used as an efficacy measure. The minimum score is 0, representing the better outcome, and the maximum value is 19, representing the worse outcome.
Time Frame: Days 1, 3, 5, 8, 11, 15, 22, and 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized with data at baseline and at each timepoint. Missing values were imputed using Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
units on a scale
  Day 3 | -0.5 (2.5) | -0.1 (2.6)
  Day 5 | -0.9 (2.8) | -0.4 (2.8)
  Day 8 | -1.5 (2.9) | -0.8 (3.3)
  Day 11 | -1.8 (3.2) | -1.1 (3.5)
  Day 15 | -2.1 (3.3) | -1.2 (3.9)
  Day 22 | -2.0 (3.8) | -1.2 (4.6)
  Day 29 | -2.2 (4.3) | -1.4 (5.0)

17. Secondary Outcome: Percentage of Participants Reporting Grade 3 and 4 Clinical and/or Laboratory Adverse Events (AEs)
Description: Grade 3 AEs are defined as events that interrupt usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Severe events are usually incapacitating. Grade 4 AEs are defined as events that are potentially life threatening.
Time Frame: Day 1 through Day 29
Population: The safety population includes all participants with available data post baseline, analyzed as treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 507 | 509
percentage of participants | 40.8 [36.5 to 45.3] | 46.8 [42.4 to 51.2]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; Test type: Superiority; Risk Difference (RD) = -6, 95% CI 2-sided [-12 to 0]

18. Secondary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs)
Description: An SAE is defined as an AE or suspected adverse reaction is considered serious if, in the view of either the investigator or the sponsor, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 29
Population: The safety population includes all participants with available data post baseline, analyzed as treated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 507 | 509
percentage of participants | 16.0 [12.9 to 19.5] | 21.0 [17.6 to 24.8]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; Test type: Superiority; Risk Difference (RD) = -5, 95% CI 2-sided [-10 to 0]

19. Secondary Outcome: Duration of Hospitalization
Description: Duration of hospitalization was determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
Days
  Including imputation for participants who died | 8 [5 to 15] | 8 [5 to 20]
  Restricted to participants who did not die: number analyzed (Participants) | 491 | 481
  Restricted to participants who did not die | 8 [5 to 13] | 8 [5 to 15]

20. Secondary Outcome: Duration of New Non-invasive Ventilation or High Flow Oxygen Use
Description: Duration of new non-invasive ventilation or high flow oxygen use was measured in days among participants who were not on non-invasive ventilation or high-flow oxygen use at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were not on non-invasive ventilation or high-flow oxygen at baseline but who subsequently required non-invasive or high-flow oxygen.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 70 | 82
Days
  Including imputations for participants who died | 6 [3 to 15] | 4.5 [2 to 11]
  Among participants who did not die: number analyzed (Participants) | 65 | 72
  Among participants who did not die | 5 [3 to 10] | 4 [2 to 7]

21. Secondary Outcome: Duration of New Oxygen Use
Description: Duration of new oxygen use was measured in days among participants who were not on oxygen at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were not on oxygen at baseline but who subsequently required oxygen.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 16 | 29
Days
  Including imputations for participants who died | 3 [2 to 4] | 3 [2 to 6]
  Among participants who did not die | 3 [2 to 4] | 3 [2 to 6]

22. Secondary Outcome: Duration of New Ventilator or Extracorporeal Membrane Oxygenation (ECMO) Use
Description: Duration of new ventilator or ECMO use was measured in days among participants who were not on a ventilator or ECMO at baseline, determined two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants not on a ventilator or ECMO at baseline but who subsequently required a ventilator or ECMO.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 46 | 70
Days
  Including imputations for participants who died | 16 [8 to 28] | 27 [12 to 28]
  Among participants who did not die: number analyzed (Participants) | 39 | 52
  Among participants who did not die | 13 [6 to 22] | 20 [10 to 27]

23. Secondary Outcome: Duration of Oxygen Use
Description: Duration of oxygen use was measured in days among participants who were on oxygen in based, calculated in two ways. The first includes imputations for participants who died. The second method is restricted to participants who did not die.
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants who were on oxygen at baseline.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 445 | 446
Days
  Including imputations for participants who died | 10 [4 to 27] | 12 [4 to 28]
  Among participants who did not die: number analyzed (Participants) | 421 | 409
  Among participants who did not die | 9 [4 to 24] | 10 [4 to 28]

24. Secondary Outcome: Percentage of Participants Discontinued or Temporarily Suspended From Investigational Therapeutics
Description: Participants may have been discontinued from investigational therapeutics due to discharge or death. The halting or slowing of the infusion for any reason was collected, as was missed doses in the series of 10 doses of Remdesivir, or in the 14 doses of Baricitinib/placebo.
Time Frame: Day 1 through Day 14
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Received less than 10 Infusions of Remdesivir due to Discharge | 55 [50 to 59] | 51 [47 to 55]
  Received less than 10 Infusions of Remdesivir due to Death | 0 [0 to 1] | 1 [0 to 2]
  Received less than 14 doses of Baricitinib/Placebo due to Discharge | 66 [62 to 70] | 59 [55 to 64]
  Received less than 14 doses of Baricitinib/Placebo due to Death | 0 [0 to 1] | 1 [1 to 3]
  Had Any Infusions of Remdesivir Halted or Slowed | 2 [1 to 4] | 2 [1 to 3]
  Had Any Oral Doses of Baricitinib/Placebo Modified | 16 [13 to 20] | 18 [14 to 21]
  Missed Any Maintenance Dose of Remdesivir | 23 [20 to 27] | 27 [23 to 31]
  Missed Any Oral Dose of Baricitinib/Placebo | 30 [26 to 34] | 34 [30 to 38]
  Terminated Early Prior to Completing 10 Infusions of Remdesivir | 3 [2 to 5] | 4 [3 to 6]
  Terminated Early Prior to Completing 14 doses of Baricitinib/Placebo | 4 [2 to 6] | 5 [3 to 7]

25. Secondary Outcome: Percentage of Participants Requiring New Ventilator or Extracorporeal Membrane Oxygenation (ECMO) Use
Description: The percentage of participants requiring new ventilator or ECMO use was determined as the percentage not on a ventilator or ECMO at baseline
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants not on a ventilator or ECMO at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 461 | 461
percentage of participants | 10 [8 to 13] | 15 [12 to 19]

26. Secondary Outcome: Percentage of Participants Requiring New Oxygen Use
Description: The percentage of participants requiring new oxygen use was determined as the percentage of participants not requiring oxygen at baseline
Time Frame: Day 1 through Day 29
Population: The analysis population is restricted to randomized participants not requiring oxygen at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 70 | 72
percentage of participants | 23 [15 to 34] | 40 [30 to 52]

27. Secondary Outcome: Mean Change in the Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. A positive change indicates a worsening and a negative change is an improvement.
Time Frame: Day 1, 3, 5, 8, 11, 15, 22, and 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized reporting a clinical score. Missing values were imputed using Last Observation Carried Forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
units on a scale
  Day 3 | 0.1 (0.5) | 0.1 (0.6)
  Day 5 | 0.0 (0.7) | 0.0 (0.7)
  Day 8 | -0.3 (0.9) | -0.1 (0.9)
  Day 11 | -0.4 (1.0) | -0.2 (1.0)
  Day 15 | -2.3 (1.9) | -1.9 (2.0)
  Day 22 | -2.7 (1.9) | -2.3 (2.1)
  Day 29 | -2.9 (1.9) | -2.5 (2.1)

28. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 15
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. Data was imputed using last observation carried forward or worst possible score based on hospitalization status (2 if not hospitalized, 7 if hospitalized) when there was a change in hospitalization status since last score. Deaths were imputed as an 8.
Time Frame: Day 15
Population: The intent-to-treat (ITT) population includes all participants who were randomized.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Death at or before study visit | 2 [1 to 4] | 3 [2 to 5]
  Hospitalized, on invasive mech. vent. or ECMO | 9 [7 to 12] | 16 [13 to 19]
  Hospitalized, on non-invasive vent./high flow O2 | 4 [3 to 6] | 4 [2 to 6]
  Hospitalized, requiring supplemental oxygen | 8 [6 to 11] | 10 [7 to 13]
  Hospitalized, not on O2, requiring ongoing care | 6 [4 to 8] | 3 [2 to 5]
  Hospitalized, not requiring O2, no longer req care | 2 [1 to 3] | 1 [0 to 2]
  Not hospitalized, limit on activities/req home O2 | 34 [30 to 39] | 31 [28 to 36]
  Not hospitalized, no limitations on activities | 34 [30 to 39] | 32 [28 to 36]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; Test type: Superiority; p = 0.44, Regression, Logistic; Odds Ratio (OR) = 1.26, 95% CI 2-sided [1.01 to 1.57]

29. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 1
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities.
Time Frame: Day 1
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Death at or before study Visit | 0 [0 to 1] | 0 [0 to 1]
  Hospitalized, on invasive mech. vent. or ECMO | 10 [8 to 13] | 11 [9 to 14]
  Hospitalized, on non-invasive vent./high flow O2 | 20 [17 to 24] | 22 [18 to 26]
  Hospitalized, requiring supplemental oxygen | 56 [52 to 60] | 53 [49 to 58]
  Hospitalized, not on O2, requiring ongoing care | 14 [11 to 17] | 14 [11 to 17]
  Hospitalized, not requiring O2, no longer req care | 0 [0 to 1] | 0 [0 to 1]
  Not hospitalized, limit on activities/req home O2 | 0 [0 to 1] | 0 [0 to 1]
  Not hospitalized, no limitations on activities | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discontinued | 0 [0 to 1] | 0 [0 to 1]

30. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 3
Description: as for outcome 29
Time Frame: Day 3
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Death at or before study Visit | 0.4 [0 to 1] | 0 [0 to 1]
  Hospitalized, on invasive mech. vent. or ECMO | 15 [12 to 18] | 16 [13 to 20]
  Hospitalized, on non-invasive vent./high flow O2 | 22 [18 to 25] | 22 [18 to 25]
  Hospitalized, requiring supplemental oxygen | 45 [41 to 50] | 44 [40 to 49]
  Hospitalized, not on O2, requiring ongoing care | 16 [13 to 20] | 14 [12 to 18]
  Hospitalized, not requiring O2, no longer req care | 0.2 [0 to 1] | 1 [0 to 2]
  Not hospitalized, limit on activities/req home O2 | 0 [0 to 1] | 0 [0 to 1]
  Not hospitalized, no limitations on activities | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 0.2 [0 to 1] | 0.4 [0 to 1]
  No clinical status score reported - Discontinued | 1 [1 to 3] | 2 [1 to 4]

31. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 5
Description: as for outcome 29
Time Frame: Day 5
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Death at or before study Visit | 1 [0 to 2] | 0 [0 to 1]
  Hospitalized, on invasive mech. vent. or ECMO | 15 [12 to 19] | 18 [15 to 21]
  Hospitalized, on non-invasive vent./high flow O2 | 17 [14 to 20] | 18 [15 to 22]
  Hospitalized, requiring supplemental oxygen | 35 [31 to 39] | 33 [29 to 37]
  Hospitalized, not on O2, requiring ongoing care | 19 [16 to 22] | 15 [12 to 18]
  Hospitalized, not requiring O2, no longer req care | 1 [0 to 2] | 1 [0 to 2]
  Not hospitalized, limit on activities/req home O2 | 0.2 [0 to 1] | 0 [0 to 1]
  Not hospitalized, no limitations on activities | 0.2 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0.2 [0 to 1]
  No clinical status score reported - Discharged | 10 [8 to 13] | 13 [10 to 16]
  No clinical status score reported - Discontinued | 2 [1 to 4] | 3 [2 to 5]

32. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 8
Description: as for outcome 29
Time Frame: Day 8
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Death at or before study Visit | 1 [0 to 2] | 1 [0 to 2]
  Hospitalized, on invasive mech. vent. or ECMO | 13 [11 to 17] | 18 [15 to 22]
  Hospitalized, on non-invasive vent./high flow O2 | 11 [8 to 14] | 12 [9 to 15]
  Hospitalized, requiring supplemental oxygen | 18 [15 to 22] | 18 [15 to 22]
  Hospitalized, not on O2, requiring ongoing care | 12 [10 to 16] | 10 [7 to 13]
  Hospitalized, not requiring O2, no longer req care | 1 [0 to 2] | 1 [0 to 2]
  Not hospitalized, limit on activities/req home O2 | 0.2 [0 to 1] | 0 [0 to 1]
  Not hospitalized, no limitations on activities | 0.4 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0.4 [0 to 1]
  No clinical status score reported - Discharged | 40 [35 to 44] | 36 [32 to 41]
  No clinical status score reported - Discontinued | 3 [2 to 5] | 4 [3 to 6]

33. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 11
Description: as for outcome 29
Time Frame: Day 11
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Death at or before study Visit | 1 [0 to 2] | 2 [1 to 4]
  Hospitalized, on invasive mech. vent. or ECMO | 11 [9 to 14] | 16 [13 to 20]
  Hospitalized, on non-invasive vent./high flow O2 | 6 [5 to 9] | 7 [5 to 9]
  Hospitalized, requiring supplemental oxygen | 12 [10 to 15] | 10 [8 to 13]
  Hospitalized, not on O2, requiring ongoing care | 9 [6 to 11] | 7 [5 to 9]
  Hospitalized, not requiring O2, no longer req care | 1 [0 to 2] | 1 [0 to 2]
  Not hospitalized, limit on activities/req home O2 | 0 [0 to 1] | 0 [0 to 1]
  Not hospitalized, no limitations on activities | 0.2 [0 to 1] | 0.2 [0 to 2]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 1 [0 to 2]
  No clinical status score reported - Discharged | 56 [52 to 60] | 52 [48 to 56]
  No clinical status score reported - Discontinued | 3 [2 to 5] | 4 [3 to 6]

34. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 22
Description: as for outcome 29
Time Frame: Day 22
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Death at or before study Visit | 4 [3 to 6] | 6 [5 to 9]
  Hospitalized, on invasive mech. vent. or ECMO | 6 [4 to 8] | 9 [7 to 12]
  Hospitalized, on non-invasive vent./high flow O2 | 3 [2 to 5] | 1 [1 to 3]
  Hospitalized, requiring supplemental oxygen | 3 [2 to 5] | 5 [3 to 7]
  Hospitalized, not on O2, requiring ongoing care | 2 [1 to 4] | 3 [1 to 4]
  Hospitalized, not requiring O2, no longer req care | 1 [1 to 3] | 0.4 [0 to 1]
  Not hospitalized, limit on activities/req home O2 | 24 [21 to 28] | 25 [21 to 29]
  Not hospitalized, no limitations on activities | 44 [40 to 49] | 37 [33 to 42]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 4 [2 to 6] | 3 [2 to 5]
  No clinical status score reported - Discontinued | 9 [6 to 11] | 10 [8 to 13]

35. Secondary Outcome: Percentage of Participants at Each Clinical Status Using Ordinal Scale at Day 29
Description: as for outcome 29
Time Frame: Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
percentage of participants
  Death at or before study Visit | 5 [3 to 7] | 7 [5 to 10]
  Hospitalized, on invasive mech. vent. or ECMO | 3 [2 to 5] | 7 [5 to 9]
  Hospitalized, on non-invasive vent./high flow O2 | 2 [1 to 3] | 1 [1 to 3]
  Hospitalized, requiring supplemental oxygen | 2 [1 to 4] | 3 [2 to 5]
  Hospitalized, not on O2, requiring ongoing care | 3 [2 to 5] | 1 [0 to 2]
  Hospitalized, not requiring O2, no longer req care | 1 [0 to 2] | 0.2 [0 to 1]
  Not hospitalized, limit on activities/req home O2 | 23 [20 to 27] | 23 [20 to 27]
  Not hospitalized, no limitations on activities | 49 [44 to 53] | 43 [39 to 47]
  No clinical status score reported - Hospitalized | 0 [0 to 1] | 0 [0 to 1]
  No clinical status score reported - Discharged | 0.4 [0 to 1] | 1 [1 to 3]
  No clinical status score reported - Discontinued | 12 [9 to 15] | 13 [10 to 16]
  No clinical status, completed study without reporting score | 0.2 [0 to 1] | 0.2 [0 to 1]

36. Secondary Outcome: 14-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 15. The proportions reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 15
Population: The ITT population consists of all participants as randomized.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
proportion of participants | 0.02 [0.01 to 0.03] | 0.03 [0.02 to 0.05]

37. Secondary Outcome: 28-day Participant Mortality
Description: The mortality rate was determined as the proportion of participants who died by study Day 29. The proportions reported are Kaplan-Meier estimates.
Time Frame: Day 1 through Day 29
Population: The ITT population includes all participants as randomized.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
proportion of participants | 0.05 [0.03 to 0.08] | 0.08 [0.06 to 0.11]

38. Secondary Outcome: Time to an Improvement of One Category Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 8) Death; 7) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5) Hospitalized, requiring supplemental oxygen; 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 3) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2) Not hospitalized, limitation on activities and/or requiring home oxygen; 1) Not hospitalized, no limitations on activities. Time to improvement by at least one category was determined for each participant
Time Frame: Day 1 through Day 29
Population: The ITT population includes all participants as randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
Days | 6.0 [5.0 to 7.0] | 8.0 [7.0 to 9.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; Test type: Superiority; p = 0.002, Log Rank; Cox Proportional Hazard = 1.21, 95% CI 2-sided [1.06 to 1.39]

39. Secondary Outcome: Time to an Improvement of Two Categories Using an Ordinal Scale
Description: The ordinal scale is an assessment of the clinical status at the first assessment of a given study day. The scale is as follows: 1) Death; 2) Hospitalized, on invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO); 3) Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4) Hospitalized, requiring supplemental oxygen; 5) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID-19 related or otherwise); 6) Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 7) Not hospitalized, limitation on activities and/or requiring home oxygen; 8) Not hospitalized, no limitations on activities. Time to improvement by at least two categories was determined for each participant
Time Frame: Day 1 through Day 29
Population: The ITT population includes all participants as randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
Days | 12.0 [12.0 to 13.0] | 13.0 [NA to NA] — Due to a large number of subjects improving 13 days post randomization there is little variability at the 50th percentile and the methodology described by Klein and Moeschberger (1997) is unable to compute a confidence interval
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; Test type: Superiority; p = 0.005, Log Rank; Cox Proportional Hazard = 1.20, 95% CI 2-sided [1.05 to 1.38]

40. Secondary Outcome: Time to Discharge or to a NEWS of 2 or Less and Maintained for 24 Hours, Whichever Occurs First
Description: The NEW score has demonstrated an ability to discriminate patients at risk of poor outcomes. This score is based on 7 clinical parameters (respiration rate, oxygen saturation, any supplemental oxygen, temperature, systolic blood pressure, heart rate, level of consciousness). The NEW Score is being used as an efficacy measure. The minimum score is 0, representing the better outcome, and the maximum value is 19, representing the worse outcome. The time to discharge or a NEWS of less than or equal to 2 was determined for each participant.
Time Frame: Day 1 through Day 29
Population: The ITT population includes participants as randomized, and restricted to those with a baseline NEWS score of 2 or greater.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 361 | 334
Days | 6.0 [6.0 to 7.0] | 7.0 [6.0 to 9.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; Test type: Superiority; p = 0.003, Log Rank; Cox Proportional Hazard = 1.24, 95% CI 2-sided [1.07 to 1.44]

41. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP)
Description: Blood to evaluate CRP was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 446 | 455
mg/L
  Day 3 | -23.035 (169.442) | -18.671 (102.661)
  Day 5: number analyzed (Participants) | 368 | 367
  Day 5 | -58.935 (110.364) | -30.908 (150.076)
  Day 8: number analyzed (Participants) | 241 | 250
  Day 8 | -78.411 (104.943) | -62.038 (125.254)
  Day 11: number analyzed (Participants) | 159 | 181
  Day 11 | -103.789 (124.751) | -88.881 (159.184)
  Day 15: number analyzed (Participants) | 221 | 240
  Day 15 | -122.339 (110.502) | -112.588 (155.762)
  Day 29: number analyzed (Participants) | 217 | 219
  Day 29 | -131.333 (115.243) | -122.342 (268.733)

42. Secondary Outcome: Change From Baseline in D-dimer Concentration
Description: Blood to evaluate d-dimer concentration was collected at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29, with the Day 1 assessment serving as baseline. Participants who had been discharged had blood collected if infection control measures allowed for in-person visits after discharge.
Time Frame: Days 1, 3, 5, 8, 11, 15 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 436 | 432
mg/L
  Day 3 | -0.374 (7.062) | 0.384 (5.663)
  Day 5: number analyzed (Participants) | 352 | 347
  Day 5 | 0.053 (10.968) | -0.149 (5.978)
  Day 8: number analyzed (Participants) | 227 | 230
  Day 8 | -0.271 (9.994) | 0.351 (5.387)
  Day 11: number analyzed (Participants) | 153 | 160
  Day 11 | 0.622 (12.779) | 0.309 (7.283)
  Day 15: number analyzed (Participants) | 215 | 230
  Day 15 | -0.988 (11.352) | -0.422 (6.579)
  Day 29: number analyzed (Participants) | 223 | 206
  Day 29 | 0.774 (27.229) | -0.219 (10.386)

43. Primary Outcome: Time to Recovery by Race
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
Days
  Asian: number analyzed (Participants) | 49 | 52
  Asian | 10 [7.0 to 13.0] | 10.0 [9.0 to 13.0]
  Black or African American: number analyzed (Participants) | 77 | 79
  Black or African American | 7.0 [5.0 to 8.0] | 6.0 [5.0 to 8.0]
  White: number analyzed (Participants) | 251 | 245
  White | 7.0 [5.0 to 8.0] | 7.0 [6.0 to 9.0]
  Other: number analyzed (Participants) | 138 | 142
  Other | 7.0 [6.0 to 8.0] | 8.0 [6.0 to 11.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; This analysis is for Asian participants; Test type: Superiority; Cox Proportional Hazard = 1.11, 95% CI 2-sided [0.73 to 1.68]
Statistical Analysis 2: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; This analysis is for Black or African American participants; Test type: Superiority; Cox Proportional Hazard = 1.06, 95% CI 2-sided [0.75 to 1.50]
Statistical Analysis 3: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; This analysis is for White participants; Test type: Superiority; Cox Proportional Hazard = 1.13, 95% CI 2-sided [0.93 to 1.37]
Statistical Analysis 4: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; This analysis is for Race of Other participants; Test type: Superiority; Cox Proportional Hazard = 1.34, 95% CI 2-sided [1.03 to 1.74]

44. Primary Outcome: Time to Recovery by Ethnicity
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized and for whom ethnicity was reported
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 509 | 508
Days
  Not Hispanic or Latino: number analyzed (Participants) | 246 | 240
  Not Hispanic or Latino | 7.0 [6.0 to 8.0] | 9.0 [7.0 to 10.0]
  Hispanic or Latino: number analyzed (Participants) | 263 | 268
  Hispanic or Latino | 7.0 [6.0 to 8.0] | 7.0 [6.0 to 9.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; This analysis is for Not Hispanic or Latino participants; Test type: Superiority; Cox Proportional Hazard = 1.31, 95% CI 2-sided [1.08 to 1.60]
Statistical Analysis 2: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; This analysis is for Hispanic or Latino participants; Test type: Superiority; Cox Proportional Hazard = 1.08, 95% CI 2-sided [0.89 to 1.31]

45. Primary Outcome: Time to Recovery by Sex
Description: as for outcome 1
Time Frame: Day 1 through Day 29
Population: The intent-to-treat (ITT) population includes all participants who were randomized
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
Number analyzed (Participants) | 515 | 518
Days
  Male: number analyzed (Participants) | 319 | 333
  Male | 7.0 [6.0 to 8.0] | 9.0 [7.0 to 11.0]
  Female: number analyzed (Participants) | 196 | 185
  Female | 7.0 [6.0 to 8.0] | 7.0 [6.0 to 7.0]
Statistical Analysis 1: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; This analysis is for Male participants; Test type: Superiority; Cox Proportional Hazard = 1.23, 95% CI 2-sided [1.04 to 1.46]
Statistical Analysis 2: Comparison: Remdesivir Plus Baricitinib vs Remdesivir Plus Placebo; This analysis is for Female participants; Test type: Superiority; Cox Proportional Hazard = 1.06, 95% CI 2-sided [0.85 to 1.32]

ADVERSE EVENTS:
Time Frame: Serious and Grade 3 and 4 non-serious adverse events were collected for 29 days after the first dose. Laboratory values were systematically assessed at Days 1, 3, 5, 8, and 11 while participants were inpatient, and at Days 15 and 29. Treatment emergent and fatal AEs are reported.
Description: Given the severity of underlying illness, participants were expected to have many symptoms and abnormalities in vital signs and laboratory values. All Grade 3 and 4 AEs were captured as AEs in this trial. Grade 2 or higher, suspected drug-related hypersensitivity reaction or deep vein thrombosis of any grade was reported as an AE in this trial. All cause mortality was calculated for the ITT population, while SAEs and AEs reflect the as treated population.
Arm/Group | Remdesivir Plus Baricitinib | Remdesivir Plus Placebo
All-Cause Mortality (participants affected / at risk) | 24/515 | 37/518
Serious Adverse Events (participants affected / at risk) | 88/507 | 109/509
Other Adverse Events (participants affected / at risk) | 147/507 | 164/509
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir Plus Baricitinib (N=507) | Remdesivir Plus Placebo (N=509)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 29 (30) | 37 (38)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 16 (16)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 11 (11)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (10)
Septic shock (Infections and infestations) | 4 (4) | 8 (8)
Hypotension (Vascular disorders) | 6 (6) | 5 (5)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7)
Pneumonia (Infections and infestations) | 2 (2) | 8 (8)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Shock (Vascular disorders) | 2 (2) | 4 (4)
Cardiac arrest (Cardiac disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Sepsis (Infections and infestations) | 2 (2) | 5 (5)
Renal failure (Renal and urinary disorders) | 0 (0) | 5 (5)
Pulseless electrical activity (Cardiac disorders) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3)
Chest pain (General disorders) | 2 (2) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Distributive shock (Vascular disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Aspergillus infection (Infections and infestations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remdesivir Plus Baricitinib (N=507) | Remdesivir Plus Placebo (N=509)
Glomerular filtration rate decreased (Investigations) | 50 (52) | 45 (46)
Hyperglycaemia (Metabolism and nutrition disorders) | 29 (34) | 40 (47)
Haemoglobin decreased (Investigations) | 30 (32) | 31 (32)
Lymphocyte count decreased (Investigations) | 25 (28) | 36 (36)
Anaemia (Blood and lymphatic system disorders) | 25 (28) | 31 (40)
Blood glucose increased (Investigations) | 26 (26) | 28 (28)
Acute kidney injury (Renal and urinary disorders) | 16 (17) | 27 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/79/NCT04401579/Prot_002.pdf
  • Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT04401579/SAP_003.pdf
  • Informed Consent Form (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT04401579/ICF_001.pdf